CLINICAL TRIAL: NCT05579912
Title: The Diagnostic Dilemma of Anastomotic Leak in Esophagogastric Surgery: Is it Safe to Feed the Patient?
Brief Title: The Diagnostic Dilemma of Anastomotic Leak in Esophagogastric Surgery
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/00612
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Anastomotic Leak
Keywords: anastomotic leak; esophagogastric surgery; bariatric surgery; anastamosis
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Esophagogastric Surgery Patients: Patients who underwent esophageal and gastric resections requiring an anastomosis from January 2001 to March 2019
  Interventions: Procedure: Esophageal and gastric resections requiring an anastomosis

INTERVENTIONS:
Procedure: Esophageal and gastric resections requiring an anastomosis — Distal gastrectomies, total gastrectomies, bariatric gastric bypasses, subtotal esophagectomies, proximal gastrectomies, palliative bypasses, and total esophagectomies.

SUMMARY:
To study the diagnostic specificity and sensitivity of various modalities used for the assessment of anastomotic leak in esophagogastric surgery and to identify the most sensitive technique. Secondarily, to propose a clinical algorithm to guide clinicians in the diagnosis of anastomotic leaks esophagogastric surgeries.

DETAILED DESCRIPTION:
Anastomotic leak in esophagogastric surgery remains a diagnostic challenge despite advances in imaging techniques. All available modalities appear to have limited sensitivities and have significant false negatives. A high index of clinical suspicion continues to be the key element in the early diagnosis of esophagogastric anastomotic leaks. The incidence of anastomotic leak in esophagogastric surgeries is reported to range from 7-20% in various studies, and it is a major complication that increases hospital stay and mortality. It is important to identify these complications early to optimize the outcomes of these patients. There has been no study till date that examines the incidence of false negative results for anastomotic leak in esophagogastric surgeries. False negative findings may give surgeons a false sense of assurance in the patient's postoperative recovery, and escalation of oral intake may result in catastrophic complications and outcomes in these patients. This study seeks to identify the most sensitive modality in the diagnosis of esophagogastric anastomotic leaks in a retrospective series of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing any of the following surgeries at National University Hospital, Singapore between January 2001 and March 2019:
* Distal gastrectomies
* Total gastrectomies
* Bariatric gastric bypasses
* Subtotal esophagectomies
* Proximal gastrectomies
* Palliative bypasses
* Total esophagectomies

Exclusion Criteria:

* Under 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing esophagogastric surgeries requiring anastamosis.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak | Surgery day
  To identify key clinical parameters that are predictive of anastomotic leak and to evaluate the effectiveness of various investigations for diagnosing anastomotic leak following upper gastrointestinal surgeries involving anastomosis

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urschel JD. Esophagogastrostomy anastomotic leaks complicating esophagectomy: a review. Am J Surg. 1995 Jun;169(6):634-40. doi: 10.1016/s0002-9610(99)80238-4. PMID 7771633
- [Background] Bruce J, Krukowski ZH, Al-Khairy G, Russell EM, Park KG. Systematic review of the definition and measurement of anastomotic leak after gastrointestinal surgery. Br J Surg. 2001 Sep;88(9):1157-68. doi: 10.1046/j.0007-1323.2001.01829.x. PMID 11531861